CLINICAL TRIAL: NCT04039113
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group, Multicenter Phase 2a Study to Explore the Efficacy and Safety of Tezepelumab in Patients With Moderate to Very Severe Chronic Obstructive Pulmonary Disease (COPD) (COURSE)
Brief Title: Tezepelumab COPD Exacerbation Study
Acronym: COURSE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5241C00001; 2019-001363-67 (EudraCT Number)
Record Dates: First submitted 2019-07-29; First posted 2019-07-31 (Actual); Results first posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; Moderate COPD; Severe COPD; chronic obstructive pulmonary disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — tezepelumab

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in a 1:1 ratio to either tezepelumab or matching placebo both administered subcutaneously.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tezepelumab (Active Comparator): Tezepelumab, SC, Q4W
  Interventions: Biological: Tezepelumab
- Matching Placebo (Placebo Comparator): Matching placebo, SC, Q4W
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Tezepelumab — Tezepelumab subcutaneous injection
  Arms: Tezepelumab
Other: Placebo — Placebo subcutaneous injection
  Arms: Matching Placebo

SUMMARY:
A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Group, Phase 2a Study to Explore the Efficacy and Safety of Tezepelumab in Adults with Moderate to Very Severe Chronic Obstructive Pulmonary Disease (COPD)

DETAILED DESCRIPTION:
This is a Phase 2a, multicenter, randomized, double-blind, placebo-controlled, parallel group study to evaluate the safety and efficacy of tezepelumab in adults with moderate to very severe chronic obstructive pulmonary disease (COPD) receiving triple inhaled maintenance therapy, and having had 2 or more documented COPD exacerbations in the 12 months prior to Visit 1. Approximately, 338 subjects will be randomized globally. Subjects will be stratified by region and prior number of exacerbations (2 vs. 3 or more). Subjects will receive tezepelumab, or placebo, administered via subcutaneous injection at the study site, over a 52 week treatment period. The study also includes a post-treatment follow-up period of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. History of moderate to very severe physician-diagnosed COPD for at least 12 months prior to enrolment with a post-bronchodilator FEV1/FVC<0.70 and a post-bronchodilator FEV1 ≥20% and ≤80% of predicted normal value.
2. History of at least 2 documented moderate to severe COPD exacerbations within 2 to 52 weeks prior to enrollment.
3. CAT score of ≥15 at enrollment and on day of randomization.
4. Documented treatment with triple therapy for COPD (medium or high dose ICS/LABA/LAMA) throughout the year prior to enrollment. The dose of ICS should be stable for 3 months prior to enrollment.

Exclusion Criteria:

1. Clinically important pulmonary disease other than COPD, as judged by the Investigator (including current or historic asthma diagnosis).
2. Any disorder, including, but not limited to, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious (including risk factors for pneumonia), endocrine, metabolic, hematological, psychiatric, or major physical impairment that is not stable.
3. Major surgery within 8 weeks before enrollment.
4. History of clinically significant infection requiring antibiotics or antiviral medication within 14 days before enrollment.
5. Pregnant or breastfeeding.
6. The chest/lungs with pathology that precludes the patient's ability to complete the study
7. The patient has active COVID 19 infection during screening period.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 337 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dave Singh, MD, Principal Investigator — Division of Infection, Immunity & Resp Medicine, The University of Manchester, United Kingdom
Locations (83):
- United States (27):
  - Research Site, Dothan, Alabama
  - Research Site, Huntington Beach, California
  - Research Site, Newport Beach, California
  - Research Site, Upland, California
  - Research Site, Westminster, California
  - Research Site, New Haven, Connecticut
  - Research Site, Brandon, Florida
  - Research Site, Orlando, Florida
  - Research Site, Panama City, Florida
  - Research Site, Tampa, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Buckley, Michigan
  - Research Site, Albuquerque, New Mexico
  - Research Site, Charlotte, North Carolina
  - Research Site, Mooresville, North Carolina
  - Research Site, New Bern, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Edmond, Oklahoma
  - Research Site, Medford, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Rock Hill, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, McKinney, Texas
  - Research Site, Abingdon, Virginia
  - Research Site, Everett, Washington
- Canada (10):
  - Research Site, Calgary, Alberta
  - Research Site, Sherwood Park, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Truro, Nova Scotia
  - Research Site, Burlington, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saint-Charles-Borromée, Quebec
  - Research Site, Trois-Rivières, Quebec
- Denmark (7):
  - Research Site, Aalborg
  - Research Site, Aarhus N
  - Research Site, Hvidovre
  - Research Site, København NV
  - Research Site, Odense C
  - Research Site, Roskilde
  - Research Site, Vejle
- France (7):
  - Research Site, Amiens
  - Research Site, Brest
  - Research Site, Grenoble
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Nantes
- Germany (5):
  - Research Site, Berlin
  - Research Site, Frankfurt
  - Research Site, Großhansdorf
  - Research Site, Lübeck
  - Research Site, Mainz
- Israel (6):
  - Research Site, Ashkelon
  - Research Site, Beersheba
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Rehovot
- Netherlands (4):
  - Research Site, Eindhoven
  - Research Site, Heerlen
  - Research Site, Rotterdam
  - Research Site, Zutphen
- South Korea (5):
  - Research Site, Daegu
  - Research Site, Incheon
  - Research Site, Jeonju
  - Research Site, Seoul
  - Research Site, Uijeongbu-si
- Spain (5):
  - Research Site, Alzira
  - Research Site, Barcelona
  - Research Site, Granada
  - Research Site, Málaga
  - Research Site, Mérida (Badajoz)
- United Kingdom (7):
  - Research Site, Bradford
  - Research Site, Chertsey
  - Research Site, Cottingham
  - Research Site, Glasgow
  - Research Site, London
  - Research Site, Newcastle upon Tyne
  - Research Site, Wakefield

REFERENCES:
- [Derived] Singh D, Brightling CE, Rabe KF, Han MK, Christenson SA, Drummond MB, Papi A, Pavord ID, Molfino NA, Almqvist G, Kotalik A, Hellqvist A, Golabek M, Sindhwani NS, Ponnarambil SS; COURSE study investigators. Efficacy and safety of tezepelumab versus placebo in adults with moderate to very severe chronic obstructive pulmonary disease (COURSE): a randomised, placebo-controlled, phase 2a trial. Lancet Respir Med. 2025 Jan;13(1):47-58. doi: 10.1016/S2213-2600(24)00324-2. Epub 2024 Dec 6. PMID 39653044
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5241C00001&attachmentIdentifier=65833b32-3e84-4701-bf38-a187adc98a98&fileName=d5241c00001-study-synopsis_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 80 centres in 10 countries. A total of 579 participants were screened of which 337 were randomised. Of the 337 randomised, 333 participants received treatment. 4 participants randomised in error and did not receive treatment. 187 participants not randomised were due to screen failures.
Pre-assignment Details: The study consisted of a screening period for approximately 6 weeks. At the end of the screening period, participants were randomised in 1:1 ratio for tezepelumab or placebo. Randomisation was stratified by region (North America, Europe, Asia), and number of prior exacerbations (2, >=3) recorded at randomisation in IWRS.
Groups:
- Tezepelumab: 420 mg Tezepelumab injection delivered subcutaneously every 4 weeks up to maximum of 52 weeks (last dose given at week 48).
- Placebo: Matching Placebo injection delivered subcutaneously every 4 weeks up to maximum of 52 weeks (last dose given at week 48).
Period: Overall Study
Arm/Group | Tezepelumab | Placebo
Started | 169 | 168
Received Treatment | 165 | 168
Completed Treatment | 138 | 138
Completed (Includes subjects who completed treatment and study, and subjects who discontinued treatment but completed study assessments up to follow up to Visit 16 (Week 52).) | 146 | 150
Not Completed | 23 | 18
Not completed — Withdrawal by Subject | 8 | 11
Not completed — Lost to Follow-up | 1 | 1
Not completed — Adverse Event | 2 | 2
Not completed — Death | 2 | 4
Not completed — Site Closure | 6 | 0
Not completed — Failure to meet randomisation criteria | 4 | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set included all participants randomised to study treatment who received at least one dose of investigational product, irrespective of their protocol adherence, and continued participation in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tezepelumab | Placebo | Total
Number analyzed (Participants) | 165 | 168 | 333
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Age (Years) | 67.4 (6.75) | 67.1 (7.24) | 67.2 (7.00)
Age, Customized [Count of Participants; unit: Participants] — Age groups in years
  Participants
    Age Group : >=40 - <65 | 52 | 61 | 113
    Age Group : >=65 - <=80 | 113 | 107 | 220
Sex: Female, Male [Count of Participants; unit: Participants]
  Sex: Female | 77 | 68 | 145
  Sex: Male | 88 | 100 | 188
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Ethnic Group: Hispanic or Latino | 7 | 3 | 10
  Ethnic Group: Not Hispanic or Latino | 158 | 165 | 323
  Ethnic Group: Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Other also includes Native Hawaiian or Other Pacific Islander and American Indian or Alaska Native categories
  Participants
    Race: White | 147 | 146 | 293
    Race: Black or African American | 2 | 2 | 4
    Race: Asian | 16 | 18 | 34
    Race: Other | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Rate of Moderate or Severe COPD Exacerbations in Participants With Moderate to Very Severe COPD.
Description: A COPD exacerbation was defined as a change in the participant's usual COPD symptoms that is beyond normal day-to-day variation, is acute in onset, lasts 2 or more days, and may warrant a change in regular medication and leads to any of the following: Use of systemic corticosteroids for at least 3 days, use of antibiotics for at least 3 days, an inpatient hospitalisation due to COPD, or results in death.
  Analysis was done using a negative binomial model with the response variable as the number of COPD exacerbations experienced during the follow-up for exacerbations. The model included covariates of treatment group, region, and number of exacerbations reported at randomisation as recorded in IWRS (2, >=3). The logarithm of the time at risk (in years) for exacerbation in the study is used as an offset variable.
Time Frame: From randomisation up to Week 52
Population: Full analysis set under the primary estimand, which comprised all participants randomised to study treatment who received at least one dose and included all observed data over the 52-week period regardless of whether participants remained on randomised treatment and regardless of whether participants switched to an alternative biologic treatment.
Measure: Least Squares Mean (90% Confidence Interval); unit: exacerbations per year
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 165 | 168
exacerbations per year | 1.75 [1.45 to 2.11] | 2.11 [1.77 to 2.53]
Statistical Analysis 1: Comparison: Tezepelumab vs Placebo; Test type: Superiority; p = 0.1042, Negative Binomial — 1-sided p-value; Rate Ratio = 0.83, 90% CI 2-sided [0.64 to 1.06]
Statistical Analysis 2: Comparison: Tezepelumab vs Placebo; Test type: Superiority; p = 0.2085, Negative Binomial — 2-sided p-value; Rate Ratio = 0.83, 95% CI 2-sided [0.61 to 1.11]

2. Secondary Outcome: Time to First Moderate/Severe COPD Exacerbation
Description: Time to first moderate/severe COPD exacerbation post-randomisation, presented as number of subjects with at least one moderate/severe COPD exacerbation.
Time Frame: From randomisation up to Week 52
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 165 | 168
Participants | 94 | 105

3. Secondary Outcome: Proportion of Participants COPD Exacerbation Free at Week 52
Description: An exacerbation event was defined as described in primary analysis. A participant was exacerbation free if they did not experience any moderate or severe exacerbations from randomisation to Week 52 (EOT).
Time Frame: From randomisation up to Week 52
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 165 | 168
Participants | 71 | 63

4. Secondary Outcome: Comparison of Annual Severe COPD Exacerbation Rates Over 52 Weeks
Description: An exacerbation was considered severe if it results in at least 1 of the following: Hospitalisation due to the COPD exacerbation (defined as a participant being admitted for ≥ 24 hours to an observation area, the emergency department, or other equivalent healthcare facility), or death related to COPD or COPD exacerbation.
Time Frame: From randomisation up to Week 52
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: exacerbations per year
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 165 | 168
exacerbations per year | 0.13 [0.07 to 0.24] | 0.25 [0.15 to 0.42]

5. Secondary Outcome: Proportion of Participants With >=1 Severe COPD Exacerbations Over 52 Weeks
Description: as for outcome 4
Time Frame: From randomisation up to Week 52
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 165 | 168
Participants | 16 | 22

6. Secondary Outcome: Time to First Severe COPD Exacerbation
Description: Time to first severe COPD exacerbation post-randomisation, presented as number of subjects with at least one severe COPD exacerbation.
Time Frame: From randomisation up to Week 52
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 165 | 168
Participants | 16 | 22

7. Secondary Outcome: Least Square (LS) Mean Difference in Change From Baseline in Pre-bronchodilator Forced Expiratory Volume in 1 (FEV1) at Week 52
Description: Pre-Bronchodilator FEV1 (L) was determined by spirometry at the clinic visit. FEV1 is defined as the volume of air exhaled from the lungs in the first second of a forced expiration.
  Change from baseline was obtained as an absolute difference between Week 52 measure and the baseline value.
  Baseline was defined as the last assessment recorded prior to the first dose of study treatment.
Time Frame: Baseline and Week 52
Population: Number of participants analyzed is the number of participants with an observation at Week 52. All participants from the Full Analysis Set with at least one change from baseline value at any post baseline visit contributes to the analyses.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 163 | 166
Liters | 0.026 (0.015) | -0.029 (0.015)

8. Secondary Outcome: Lease Square (LS) Mean Difference in Change From Baseline in St. George's Respiratory Questionnaire (SGRQ) Total Score at Week 52
Description: The SGRQ is a 50-item PRO instrument to measure the health status of participants with airway obstruction diseases. The total score indicates the impact of disease on overall health status. This total score is expressed as a percentage of overall impairment, in which 100 represents the worst possible health status and 0 indicates the best possible health status.
  Baseline is the measurement recorded at Week 0 (Visit 3).
Time Frame: Baseline and Week 52
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 157 | 156
units on a scale | -4.796 (1.176) | -1.863 (1.189)

9. Secondary Outcome: Proportion of Participants Achieving a Minimum Clinically Important Difference of 4 Units or More in St. George's Respiratory Questionnaire (SGRQ) Total Score at Week 52
Description: The SGRQ is a 50-item PRO instrument to measure the health status of participants with airway obstruction diseases. The total score indicates the impact of disease on overall health status. This total score is expressed as a percentage of overall impairment, in which 100 represents the worst possible health status and 0 indicates the best possible health status.
  A responder was defined as an individual who had "improvement" at Week 52 (>=4 point decrease in SGRQ total score).
Time Frame: Baseline and Week 52
Population: Number of participants analyzed is the number of participants from the Full Analysis Set with a baseline SGRQ score.
Measure: Count of Participants; unit: Participants
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 163 | 163
Participants | 65 | 59

10. Secondary Outcome: Least Square (LS) Mean Difference in Change From Baseline in COPD Assessment Tool (CAT) Total Score at Week 52
Description: The CAT is an 8-item PRO developed to measure the impact of COPD on health status. A CAT total score is the sum of item responses. Scores range from 0-40 with higher scores indicative of greater COPD impact on health status.
  Baseline was defined as the value at the randomisation visit (Visit 3). If the Visit 3 measurement was missing, the screening value was used as baseline instead.
Time Frame: Baseline and Week 52
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 159 | 162
units on a scale | -3.037 (0.524) | -1.182 (0.524)

11. Secondary Outcome: Serum Concentration of Tezepelumab
Description: Blood samples were collected to determine the serum concentration of Tezepelumab.
  With the exception of Week 0 and Week 64, only pre-dose data from samples collected between 21 and 35 days after previous dose of investigational product were included.
Time Frame: Pre-dose at weeks 0, 4, 12, 24, 36 and also at weeks 52 and 64 where no dosing was scheduled
Population: The Pharmacokinetic (PK) analysis set comprises all subjects who received at least one dose of tezepelumab and have at least one detectable serum concentration post first dose that is not affected by factors such as protocol deviations (e.g. disallowed medication or incorrect study medication received).
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mg/mL)
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 162 | 0
microgram per milliliter (mg/mL)
  Week 0 | NA (NA) — Below the lower limit of quantification (LLOQ). The LLOQ is 0.010 micrograms per milliliter. |
  Week 4: number analyzed (Participants) | 151 | 0
  Week 4 | 25.881 (11.8828) |
  Week 12: number analyzed (Participants) | 127 | 0
  Week 12 | 44.316 (19.0716) |
  Week 24: number analyzed (Participants) | 129 | 0
  Week 24 | 49.093 (21.2414) |
  Week 36: number analyzed (Participants) | 118 | 0
  Week 36 | 48.667 (22.2241) |
  Week 52: number analyzed (Participants) | 109 | 0
  Week 52 | 52.659 (26.1703) |
  Follow-up Week 64: number analyzed (Participants) | 129 | 0
  Follow-up Week 64 | 6.602 (6.1832) |

12. Secondary Outcome: Number of Participants With Anti-Drug Antibody (ADA) Response to Tezepelumab
Description: Blood samples were measured for the presence of ADAs for tezepelumab using validated assays. Treatment-induced ADA positive was defined as ADA negative at baseline and post-baseline ADA positive. Treatment-boosted ADA positive was defined as baseline positive ADA titre that was boosted to a 4 fold or higher level following IP administration. TE-ADA positive was defined as the sum of treatment-induced ADA positive and treatment-boosted ADA positive. ADA incidence is the proportion of TE-ADA positive subjects in a population. ADA persistently positive was defined as ADA positive at >= 2 post-baseline assessments or ADA positive at last post-baseline assessment. ADA transiently positive was defined as having at least one post-baseline ADA positive assessment and not fulfilling the conditions of ADA persistently positive. Treatment-induced nAb positive was defined as nAb negative or ADA negative at baseline and nAb positive at any post-baseline visit.
Time Frame: Pre-dose at weeks 0, 4, 12, 24, 36 and also at weeks 52 and 64 where no dosing was scheduled
Population: The safety analysis set included all subjects who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 165 | 168
Participants
  ADA positive at baseline and/or post-baseline (ADA prevalence) | 10 | 19
  Any baseline ADA positive: number analyzed (Participants) | 162 | 162
  Any baseline ADA positive | 5 | 8
  Only baseline ADA positive: number analyzed (Participants) | 162 | 162
  Only baseline ADA positive | 2 | 1
  Any post-baseline ADA positive: number analyzed (Participants) | 163 | 166
  Any post-baseline ADA positive | 8 | 18
  Both baseline and at least one post-baseline ADA positive: number analyzed (Participants) | 160 | 160
  Both baseline and at least one post-baseline ADA positive | 3 | 7
  Treatment-induced ADA positive: number analyzed (Participants) | 160 | 160
  Treatment-induced ADA positive | 5 | 11
  Treatment-boosted ADA positive: number analyzed (Participants) | 160 | 160
  Treatment-boosted ADA positive | 0 | 0
  TE-ADA positive (ADA incidence): number analyzed (Participants) | 160 | 160
  TE-ADA positive (ADA incidence) | 5 | 11
  ADA persistently positive: number analyzed (Participants) | 163 | 166
  ADA persistently positive | 5 | 15
  ADA transiently positive: number analyzed (Participants) | 163 | 166
  ADA transiently positive | 3 | 3
  nAb positive at baseline and/or post-baseline (nAb prevalence) | 0 | 0
  Treatment-induced nAb positive (nAb incidence): number analyzed (Participants) | 160 | 160
  Treatment-induced nAb positive (nAb incidence) | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug until end of study at Week 64.
Description: All AE data is based off the Safety Analysis Set, which includes all subjects who received at least one dose of study treatment.
Groups:
- Teze 420 mg Q4W: 420 mg Tezepelumab injection delivered subcutaneously every 4 weeks up to maximum of 52 weeks (last dose given at week 48).
Arm/Group | Teze 420 mg Q4W | Placebo
All-Cause Mortality (participants affected / at risk) | 3/165 | 6/168
Serious Adverse Events (participants affected / at risk) | 56/165 | 58/168
Other Adverse Events (participants affected / at risk) | 78/165 | 56/168
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teze 420 mg Q4W (N=165) | Placebo (N=168)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (2)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Vascular stent stenosis (General disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatitis alcoholic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2) | 3 (3)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Diverticulitis (Infections and infestations) | 2 (2) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Meningitis viral (Infections and infestations) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 7 (7) | 5 (5)
Pneumonia bacterial (Infections and infestations) | 3 (3) | 3 (4)
Pneumonia klebsiella (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia mycoplasmal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia pseudomonal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1)
Pseudomonas bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (2)
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural dizziness (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung carcinoma cell type unspecified stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal squamous cell carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal artery occlusion (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 20 (27) | 26 (39)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Coeliac artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Iliac artery dissection (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Alcoholic pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teze 420 mg Q4W (N=165) | Placebo (N=168)
Oedema peripheral (General disorders) | 11 (11) | 8 (8)
COVID-19 (Infections and infestations) | 25 (26) | 16 (17)
Nasopharyngitis (Infections and infestations) | 17 (18) | 9 (9)
Urinary tract infection (Infections and infestations) | 5 (6) | 10 (12)
Contusion (Injury, poisoning and procedural complications) | 10 (11) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 11 (12) | 10 (12)
Dizziness (Nervous system disorders) | 9 (11) | 1 (1)
Headache (Nervous system disorders) | 3 (4) | 10 (24)
Hypertension (Vascular disorders) | 12 (13) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 9 (10) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator agrees to submit all manuscripts or abstracts to the sponsor before submission. This allows the sponsor to protect proprietary information and to provide comments.

DOCUMENTS (2):
  • Study Protocol (2022-10-18): https://cdn.clinicaltrials.gov/large-docs/13/NCT04039113/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-28): https://cdn.clinicaltrials.gov/large-docs/13/NCT04039113/SAP_001.pdf